CLINICAL TRIAL: NCT02136030
Title: A Randomized Study to Evaluate the Safety and Efficacy of Liposomal Amphotericin B and Amphotericin B Deoxycholate With or Without Flucytosine Followed by Fluconazole, for the Treatment of Cryptococcal Meningitis
Brief Title: Liposomal Amphotericin B for the Treatment of Cryptococcal Meningitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: TTY Biopharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTYLA0701
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2010-10

CONDITIONS: Cryptococcal Meningitis
Keywords: Cryptococcal meningitis
MeSH Terms: conditions — Meningitis, Cryptococcal | interventions — liposomal amphotericin B; amphotericin B, deoxycholate drug combination; Amphotericin B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lipo-AB (Experimental)
  Interventions: Drug: Liposomal amphotericin B
- Amphotericin B (Active Comparator)
  Interventions: Drug: Amphotericin B-deoxycholate

INTERVENTIONS:
Drug: Liposomal amphotericin B — 4mg/kg/day, IV infusion
  Other Names: Lipo-AB
  Arms: Lipo-AB
Drug: Amphotericin B-deoxycholate — 1mg/kg/day, IV infusion
  Other Names: Amphotericin B
  Arms: Amphotericin B

SUMMARY:
To evaluate the safety and efficacy of liposomal amphotericin B and amphotericin B deoxycholate with or without flucytosine followed by fluconazole for the treatment of cryptococcal meningitis.

DETAILED DESCRIPTION:
Subjects who meet all eligible requirements will be randomized into study group （Lipo-AB）or control group（Amphotericin B deoxycholate） in 2:1 ratio. Subjects will be treated with induction therapy in study group or in control group with flucytosine for at least 14 days, and followed by consolidation therapy for another 56 days after CSF sterilization.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with age of at least 18 years.
2. Within 7 days prior to, or at the time of screening visit, patient with cryptococcus meningitis, diagnosed by :

   1. CSF India ink staining positive OR
   2. CSF cryptococcal antigen test positive OR
   3. CSF culture positive
3. Patient or his/her legally acceptable representative has signed the written informed consent form.

Exclusion Criteria:

1. Patients have laboratory abnormalities within 3 days prior to screening visit :

   1. ALT > 5x UNL,
   2. AST > 5x UNL,
   3. Creatinine > 2mg/dl
2. Patient is pregnant or lactating.
3. Patient participate other investigational drug trial within 1 month before entering this study.
4. Patient has some indications that another systemic antifungal drug would be needed in addition to assigned drugs in study.
5. Patient had contraindication of amphotericin B or azole.
6. Patient is not available for lumbar puncture.
7. Patient with life expectancy less than 5 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2011-02; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
suscceful response rate | Day 14
  Successful response was defined as both satisfactory clinical and microbiological response at the completion of 14 days treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Yee-chun Chen, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Perfect JR, Dismukes WE, Dromer F, Goldman DL, Graybill JR, Hamill RJ, Harrison TS, Larsen RA, Lortholary O, Nguyen MH, Pappas PG, Powderly WG, Singh N, Sobel JD, Sorrell TC. Clinical practice guidelines for the management of cryptococcal disease: 2010 update by the infectious diseases society of america. Clin Infect Dis. 2010 Feb 1;50(3):291-322. doi: 10.1086/649858. PMID 20047480
- [Derived] Adler-Moore JP, Gangneux JP, Pappas PG. Comparison between liposomal formulations of amphotericin B. Med Mycol. 2016 Mar;54(3):223-31. doi: 10.1093/mmy/myv111. Epub 2016 Jan 14. PMID 26768369
- See also: Clinical trials network in Taiwan — http://www.google.com/search?q=emome&ie=utf-8&oe=utf-8